CLINICAL TRIAL: NCT04119063
Title: Evaluating Wearable Robotic Assistance on Gait Mechanics and Energetics in Individuals With Neurological Impairment
Brief Title: Evaluating Wearable Robotic Assistance on Gait
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northern Arizona University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Zachary Lerner, Principal Investigator, Northern Arizona University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 986744; 1R15HD099664-01 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: Feasibility assessment of powered orthosis assistance and resistance during walking. All participants received high frequency gait training followed by a washout period then low frequency gait training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Gait Training with Exoskeleton Assistance (Experimental): Gait training with ankle exoskeleton assistance. All participants received high frequency gait training followed by a washout period then low frequency gait training.
  Interventions: Device: powered orthosis

INTERVENTIONS:
Device: powered orthosis — Novel powered leg brace to provide assistance during walking.
  Other Names: exoskeleton

SUMMARY:
The overarching goal of this study is to improve mobility in individuals with movement disorders through advances in wearable assistance (i.e. powered orthoses).

DETAILED DESCRIPTION:
Individuals with cerebral palsy completed high frequency over-ground gait training (4x/week for 1 week) with ankle exoskeleton assistance, and then, after a 1 year washout period, the same participants will complete low frequency over-ground gait training (2x/week for 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 35 years old, inclusive.
* Either a healthy volunteer or a diagnosis of a neurologically-based walking disorder due to stroke, spinal cord injury, Parkinson's disease, or cerebral palsy.
* Must be able to understand and follow simple directions based on parent report and clinical observation during the history and physical examination.
* Able to provide verbal assent, if appropriate. If the participant is non-verbal, parental interpretation of gesticulation for assent will be used.
* The ability to read and understand English.
* Able to walk at least 30 feet with or without a walking aid (GMFCS Level I-III for individuals with cerebral palsy)

Exclusion Criteria:

• Any neurological, musculoskeletal or cardiorespiratory injury, health condition ( including pregnancy), or diagnosis other than stroke, spinal cord injury, Parkinson's disease or cerebral palsy that would affect the ability to walk as directed for short periods of time.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Orekhov G, Fang Y, Cuddeback CF, Lerner ZF. Usability and performance validation of an ultra-lightweight and versatile untethered robotic ankle exoskeleton. J Neuroeng Rehabil. 2021 Nov 10;18(1):163. doi: 10.1186/s12984-021-00954-9. PMID 34758857

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants first completed higher frequency gait training followed by a washout period and then lower frequency gait training.
Groups:
- Gait Training With Exoskeleton Assistance: All participants received high frequency gait training followed by a washout period then low frequency gait training
Period: Overall Study
Arm/Group | Gait Training With Exoskeleton Assistance
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Exoskeleton Assistance: Gait training with exoskeleton assistance at higher and lower frequencies.
  powered orthosis: Novel powered leg brace to provide assistance during walking.
Arm/Group | Exoskeleton Assistance
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: The Metabolic Energy Required to Walk
Description: The change in the metabolic energy required to walk will be measured using a portable metabolic measurement system (Cosmed K5). Units: change in % difference post vs pre gait training.
Time Frame: Measured at the pre (day 1) and post (day 4) gait training assessments
Measure: Mean (Standard Deviation); unit: % change pre vs post gait training
Groups:
- Exoskeleton Gait Training High Frequency: Gait training with ankle exoskeleton assistance at the higher frequency.
- Exoskeleton Gait Training Low Frequency: Gait training with ankle exoskeleton assistance at the lower frequency.
Arm/Group | Exoskeleton Gait Training High Frequency | Exoskeleton Gait Training Low Frequency
Number analyzed (Participants) | 6 | 6
% change pre vs post gait training | 2.42 (16.87) | -2.14 (10.59)
Statistical Analysis 1: Comparison: Exoskeleton Gait Training High Frequency vs Exoskeleton Gait Training Low Frequency; Test type: Other — Paired t-tests comparing change in % difference following high vs low frequency gait training; p = 0.204, t-test, 2 sided

2. Primary Outcome: Change in Walking Speed
Description: The change in the walking speed will be measured over-ground using a stop watch. Units: % change between post vs pre assessments
Time Frame: Measured at the pre (day 1) and post (day 4) gait training assessments
Measure: Mean (Standard Deviation); unit: % change post vs pre training
Groups:
- Gait Training With Exoskeleton Assistance High Frequency: Gait training with ankle exoskeleton assistance at the higher frequency.
- Gait Training With Exoskeleton Assistance Low Frequency: Gait training with ankle exoskeleton assistance at the lower frequency.
Arm/Group | Gait Training With Exoskeleton Assistance High Frequency | Gait Training With Exoskeleton Assistance Low Frequency
Number analyzed (Participants) | 6 | 6
% change post vs pre training | 25.39 (14.65) | 8.09 (7.10)
Statistical Analysis 1: Comparison: Gait Training With Exoskeleton Assistance High Frequency vs Gait Training With Exoskeleton Assistance Low Frequency; Test type: Other — Paired t-test; p = 0.049, t-test, 2 sided

3. Secondary Outcome: Change in Stride Length
Description: The change in the stride length will be measured by dividing the number of steps by distance traveled. Units: % change between post vs pre assessments.
Time Frame: Measured at the pre (day 1) and post (day 4) gait training assessments
Measure: Mean (Standard Deviation); unit: % change post vs pre training
Arm/Group | Gait Training With Exoskeleton Assistance High Frequency | Gait Training With Exoskeleton Assistance Low Frequency
Number analyzed (Participants) | 6 | 6
% change post vs pre training | 16.28 (9.90) | 3.87 (5.00)
Statistical Analysis 1: Comparison: Gait Training With Exoskeleton Assistance High Frequency vs Gait Training With Exoskeleton Assistance Low Frequency; Test type: Other — Paired t-tests comparing change in % difference following high vs low frequency gait training; p = 0.039, t-test, 2 sided

4. Secondary Outcome: Change in Cadence
Description: The change in the number of steps taken per minute will be measured using a counter. Units: % change between post vs pre assessments.
Time Frame: Measured at the pre (day 1) and post (day 4) gait training assessments
Measure: Mean (Standard Deviation); unit: % change post vs pre training
Arm/Group | Gait Training With Exoskeleton Assistance High Frequency | Gait Training With Exoskeleton Assistance Low Frequency
Number analyzed (Participants) | 6 | 6
% change post vs pre training | 22.47 (35.18) | 4.04 (3.32)
Statistical Analysis 1: Comparison: Gait Training With Exoskeleton Assistance High Frequency vs Gait Training With Exoskeleton Assistance Low Frequency; Test type: Other — Paired t-tests comparing change in % difference following high vs low frequency gait training; p = 0.242, t-test, 2 sided

5. Secondary Outcome: Change in Muscle Activity Variance Ratio
Description: The change in the muscle activity variance ratio of the soleus during walking will be measured using electromyography electrodes. Units: % change between post vs pre assessments.
Time Frame: Measured at the pre (day 1) and post (day 4) gait training assessments
Measure: Mean (Standard Deviation); unit: % change post vs pre training
Arm/Group | Gait Training With Exoskeleton Assistance High Frequency | Gait Training With Exoskeleton Assistance Low Frequency
Number analyzed (Participants) | 6 | 6
% change post vs pre training | -47.24 (17.44) | 18.80 (29.97)
Statistical Analysis 1: Comparison: Gait Training With Exoskeleton Assistance High Frequency vs Gait Training With Exoskeleton Assistance Low Frequency; Test type: Other — Paired t-tests comparing change in % difference following high vs low frequency gait training; p = .014, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Over the duration of the protocol, an average of two weeks.
Arm/Group | Gait Training With Exoskeleton Assistance High Frequency | Gait Training With Exoskeleton Assistance Low Frequency
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Small sample size due to participant recruitment challenges in our location and resulting from Covid 19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT04119063/Prot_SAP_000.pdf